CLINICAL TRIAL: NCT00730197
Title: Single-Dose Fasting Bioequivalence Study of Nisoldipine Extended-Release Tablets(40 mg; Mylan) and Sular® Extended Release Tablets (40 mg; First Horizon) in Healthy Volunteers
Brief Title: Fasting Bioequivalence Study of Nisoldipine Extended-Release Tablets 40 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Will Sullvan, Global Head of Product Risk and Safety Management, Mylan Inc.
Organization: MylanPharma (Unknown)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: NISO-0701
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 2008-08

CONDITIONS: Healthy

ARMS (2):
- 1 (Experimental): NISOLDIPINE EXTENDED-RELEASE TABLETS, 40 MG
  Interventions: Drug: Albuterol Sulfate Extended-Release Tablets 8 mg
- 2 (Active Comparator): Sular® Extended Release 40 mg tablets
  Interventions: Drug: VoSpire® ER Tablets 8 mg

INTERVENTIONS:
Drug: Albuterol Sulfate Extended-Release Tablets 8 mg — 8mg, single dose fed
  Arms: 1
Drug: VoSpire® ER Tablets 8 mg — 8mg, single dose fed
  Arms: 2

SUMMARY:
The objective of this study was to investigate the bioequivalence of nisoldipine extended-release 40 mg tablets (by Mylan Pharmaceuticals Inc.) with Sular® Extended-Release 40 mg tablet (manufactured for First Horizon) following a single, oral 40 mg (1 × 40 mg tablet) dose administration in healthy adult subjects under fasting conditions.

ELIGIBILITY:
I. Inclusion Criteria:

Subjects who met the following criteria were included in the study.

1. Age: 18 years and older.
2. Sex: Male and/or non-pregnant, non-lactating female.

   1. Women of childbearing potential had a negative serum beta human chorionic gonadotropin (β-HCG) pregnancy test performed within 21 days prior to the start of the study and on the evening prior to each dose administration. An additional serum (β-HCG) pregnancy test was performed upon completion of the study.
   2. Women of childbearing potential were required to practice abstinence or use an acceptable form of contraception throughout the duration of the study. No hormonal contraceptives or hormonal replacement therapies were permitted in this study. Acceptable forms of contraception included the following:

      1. intrauterine device in place for at least 3 months prior to the start of the study and remaining in place during the study period, or
      2. barrier methods containing or used in conjunction with a spermicidal agent, or
      3. surgical sterilization (tubal ligation, oophorectomy or hysterectomy) or postmenopausal accompanied with a documented postmenopausal course of at least one year.
   3. Women were not considered of childbearing potential if one of the following was reported and documented on the medical history:

      1. postmenopausal with an absence of menses for at least one (1) year, or
      2. bilateral oophorectomy with or without a hysterectomy and an absence of bleeding for at least 6 months, or
      3. total hysterectomy
   4. During the course of the study, from study screen until study exit - including the washout period, all men and women of childbearing potential must use a spermicide containing barrier method of contraception in addition to their current contraceptive method.
3. Weight: At least 60 kg (132 lbs) for men and 48 kg (106 lbs) for women with all subjects having a Body Mass Index (BMI) less than or equal to 30 but greater than or equal to 19.
4. All subjects were judged normal and healthy during a pre-study medical evaluation, (physical examination, laboratory evaluation, Hepatitis B and Hepatitis C tests, HIV test, 12-lead ECG, and urine drug screen including amphetamine, barbiturates, benzodiazepines, cannabinoid, cocaine, opiates, phencyclidine, and methadone) performed within 21 days of the initial dose of study medication.

II. Exclusion Criteria:

Subjects who met any of the following criteria were excluded from the study:

1. Institutionalized subjects were not used.
2. Social Habits:

   1. Use of any tobacco-containing products within 1 year prior to dosing.
   2. Ingestion of any alcoholic, caffeine- or xanthine-containing food or beverage within the 48 hours prior to the initial dose of study medication.
   3. Ingestion of any vitamins or herbal products within 7 days prior to the initial dose of the study medication.
   4. Any recent, significant change in dietary or exercise habits.
   5. A positive test for any drug included in the urine drug screen.
   6. History of drug and/or alcohol abuse.
3. Medications:

   1. Use of any prescription or over-the-counter (OTC) medications within the 14 days prior to the initial dose of study medication.
   2. Use of any hormonal contraceptives or hormone replacement therapy within 3 months prior to study medication dosing.
   3. Use of any medication known to alter hepatic enzyme activity within 28 days prior to the initial dose of study medication.
4. Diseases:

   1. History of any significant cardiovascular, hepatic, renal, pulmonary, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, or neurologic disease.
   2. Acute illness at the time of either the pre-study medical evaluation or dosing.
   3. A positive HIV, hepatitis B, or hepatitis C test.
5. Abnormal and clinically significant laboratory test results:

   1. Clinically significant deviation from the Guide to Clinically Relevant Abnormalities
   2. Abnormal and clinically relevant ECG tracing.
6. Donation or loss of a significant volume of blood or plasma (> 450 mL) within 28 days prior to the initial dose of study medication.
7. Subjects who have received an investigational drug within 30 days prior to the initial dose of study medication.
8. Allergy or hypersensitivity to nisoldipine, any of the inactive ingredients, or other calcium channel blocker products.
9. History of difficulties in swallowing, or any gastrointestinal disease which could affect the drug absorption.
10. Consumption of grapefruit or grapefruit containing products within 7 days of drug administration.
11. Average sitting pulse rate less than 55 beats per minute after a five minute rest at screening or prior to Period I Day 1 dosing. Pulse rate measurements were taken in triplicate with at least two (2) minutes elapsed in-between readings.
12. Average sitting systolic blood pressure less than 90 mmHg or average sitting diastolic blood pressure less than 60 mmHg following a five (5) minute rest at screening or prior to Period I Day 1 dosing. Blood pressure measurements were taken in triplicate with at least two (2) minutes elapsed in-between readings.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-02; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: James Carlson, Pharm. D., Principal Investigator — PRACS Institute Ltd.
Locations (1):
- PRACS Institute, Ltd., Fargo, North Dakota, United States

REFERENCES:
- See also: Mylan Pharmaceuticals Inc. - Clinical Trial Results — http://www.mpibiostudies.com
- See also: Daily Med - posting of most recent submitted labelling to the Food and Drug Administration (FDA) and currently in use — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html